CLINICAL TRIAL: NCT02148627
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3041658 in Healthy Subjects
Brief Title: Safety Study of LY3041658 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15164; I7P-MC-DSAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: antibody; autoimmune

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3041658 (IV) (Experimental): Single dose of LY3041658, administered as a slow intravenous (IV) infusion in escalating dose cohorts.
  Interventions: Drug: LY3041658 (IV)
- LY3041658 (SC) (Experimental): Single dose of LY3041658 administered subcutaneously (SC).
  Interventions: Drug: LY3041658 (SC)
- Placebo (Placebo Comparator): Single dose of placebo (0.9% sodium chloride injection) administered as a slow IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3041658 (SC) — Administered SC
  Arms: LY3041658 (SC)
Drug: LY3041658 (IV) — Administered as slow IV infusion
  Arms: LY3041658 (IV)
Drug: Placebo — Administered as slow IV infusion
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety of LY3041658 in healthy participants, including first generation Japanese. The study will also investigate how the drug is processed and affects key immune cells. Study participation will last 4 months.

Protocol amended in January, 2016 to include first generation Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* All:

  * Body mass index (BMI) between 18.0 to 32.0 kilogram per square meter (kg/m²).
  * Absolute neutrophil count at screening should be ≥1.8 and ≤7.2 x 10^3/microliter (uL), inclusive.
* First-generation Japanese:

  * Participant, biological parents, and biological grandparents must be of exclusive Japanese descent and born in Japan.
  * Are 20 to 65 years of age, inclusive, at the time of initial screening.

Exclusion Criteria:

- Have received antibody-based biologic agents (marketed or investigational) within 3 months or 5 half lives (t1/2) of the drug (whichever is longer) prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-06-16 (Actual); Primary Completion 2017-02-11 (Actual); Study Completion 2017-02-11 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with One or More Drug-Related Adverse Events | Baseline to study completion (Day 85)

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY3041658 | Predose through Day 85, at specified timepoints
Pharmacokinetics: Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to Time of Last Measurable Concentration (tlast) | Predose through Day 85, at specified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - PAREXEL-Phase 1 Baltimore Harbor Hospital Center, Baltimore, Maryland